CLINICAL TRIAL: NCT07246980
Title: Continuous Observational Monitoring Program for Allay™ Hydrogel Cap Safety and Success (COMPASS) Study: An Open Label Registry Study to Assess the Safety and Performance of the Allay™ Hydrogel Cap
Brief Title: Continuous Observational Monitoring Program for Allay™ Hydrogel Cap Safety and Success Study
Acronym: COMPASS
Status: Not yet recruiting | Type: Observational
Sponsor: Tulavi Therapeutics,Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0002
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Nerve Cap — Patients who have or will receive allay Hydrogel Cap

SUMMARY:
is is a multi-center, open-label, observational registry study (both prospective and retrospective) designed to evaluate the safety and performance of the allay™ Hydrogel Cap. This cap is an in situ forming implantable hydrogel medical device used in various peripheral nerve surgeries, including amputation and neuroma excision.

The study aims to gather demographic, operative, and clinical outcomes data from patients who have received the device.

The primary endpoints focus on the device's clinical performance, assessed using patient-reported outcomes (PROs). These include tracking changes in pain scores, pain intolerance, and cold intolerance, as well as the incidence of neuroma recurrence and changes in pain medication use from baseline.

Secondary endpoints concentrate on safety, monitoring the incidence of device failures, surgical complications, unplanned re-operations, and unexpected adverse device events (UADEs) within the study population. Essentially, the registry is collecting real-world data to determine how well and how safely the allay™ cap performs in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have or will receive allay™ Hydrogel Cap

Exclusion Criteria:

* Patients who have not received allay™ Hydrogel Cap

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received or will be receiving allay™ Hydrogel Cap at a participating study site are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in Pain Scores from baseline using VAS | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 month and 24 month (Post Surgery)
  Pain scores will be collected using either of the following scales:
  1) The Visual Analog Scale (VAS) or 2) The Numerical Rating Scale (NRS)
  The VAS for pain is a simple, validated tool used to measure a patient's perceived pain intensity. It consists of a straight 100 mm horizontal line labeled from "no pain" (0) on the left to "worst imaginable pain" (100) on the right. Patients are asked to mark a point on the line that corresponds to their current level of pain, which is then measured in millimeters from the zero point to quantify the score. The VAS is widely used in both clinical and research settings due to its ease of use and sensitivity to changes in pain over time.
Assessment of change in Pain scores from baseline using Numerical Rating Scale | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 month and 24 month (Post Surgery)
  The NRS is a validated pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable. The patient selects the single whole number that best reflects how severe their current pain is to them.
Assessment of change in Pain Interference from baseline using PROMIS PI Short Form 5b | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 month and 24 month (Post Surgery)
  The Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS-PI) scale is a validated tool used to assess the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. It measures the impact of pain over the past seven days using a series of standardized questions rated on a 5-point Likert scale. Scores are converted to T-scores, with higher scores indicating greater pain interference. The PROMIS-PI is widely used in clinical research due to its reliability, responsiveness, and ability to compare results across diverse patient populations.
Assessment of change in Neuropathic Pain Quality from baseline using Patient-Reported Outcome Measurement Information System (PROMIS) v2.0 Neuropathic Pain Quality 5a | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 month and 24 month (Post Surgery)
  The Patient-Reported Outcome Measurement Information System (PROMIS) v2.0 Neuropathic Pain Quality 5a is a 5-item, self-administered questionnaire for participants to assess qualities of neuropathic pain, like "numb," "tingly," and "shooting," over the past seven(7) days. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores indicate more severe neuropathic pain. It helps to accurately screen for neuropathic pain, which arises from nerve damage, versus nociceptive pain, which comes from tissue injury, and can then assess the severity of the condition.
Assessment of change in Cold Intolerance from baseline using Cold Intolerance Symptom Severity (CISS) score | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 month and 24 month (Post Surgery)
  The Cold Intolerance Symptom Severity (CISS) score is a validated patient-reported outcome measure used to assess the severity of cold intolerance, often following peripheral nerve injury or extremity trauma. The questionnaire includes six items evaluating symptoms such as pain, numbness, stiffness, color changes, and the impact on daily activities in response to cold exposure. Each item is scored on a Likert scale, with the total score ranging from 4 to 100, where higher scores indicate greater symptom severity. The CISS is commonly used in clinical research to quantify cold intolerance and monitor changes over time or in response to interventions.
Assessment of change from baseline in the average quantity of pain medication taken via the Medication Quantification Scale (MQS) at 12 months. | Baseline (Pre Surgery ), 2 Weeks, 1 month, 4 month, 12 months (Post Surgery)
  A pain medication log will be provided to each participant to complete at all visits.
  For opioid and non-opioid pain medications, the Medication Quantification Scale (MQS) Version III is a validated tool used to quantify the complexity and detriment of pain medication regimens. It calculates a single numeric value by combining medication detriment weights (ranging from 1.1 to 4.5) with dosage levels (scaled from 1 for subtherapeutic use to 4 for supratherapeutic use). A higher MQS score indicates greater potential medication detriment and/or dosage intensity. At 12 months, the study assessed changes from baseline in patients' average MQS scores.

SECONDARY OUTCOMES:
Incidence of Device Failures surgical & medical complications, unplanned re-operations, and unexpected adverse device events (UADEs) | Upto 2 years Post Surgery
  Secondary endpoints of the study include safety assessment based on the incidence of device failures, surgical & medical complications, unplanned re-operations, and unexpected adverse device events (UADEs) in the study population.

IPD SHARING:
Plan to Share IPD: Undecided